CLINICAL TRIAL: NCT05988463
Title: A Dose-Escalation Study Evaluating the Safety and Tolerability of Artesunate in Participants With Idiopathic Pulmonary Fibrosis (SAFE-IPF)
Brief Title: Dose-Escalation Study of Artesunate Patients With IPF
Acronym: SAFE-IPF
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph C. Wu (Other)
Responsible Party: Sponsor-Investigator, Joseph C. Wu, Director, Stanford Cardiovascular Institute, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 71488
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: shortness of breath, fibrosis, cough, hypoxemia
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Dyspnea; Fibrosis; Cough; Hypoxia

STUDY DESIGN:
Intervention Model Description: RAndomized double blind label, dose escalation treatment study
Masking Description: Randomization and masking will be done via a medical software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Artesunate (Experimental): Experimental group
  Interventions: Drug: Artesuante; Other: Placebo capsules
- Placebo (No Intervention): Control

INTERVENTIONS:
Drug: Artesuante — Artesunate capsules administered orally twice daily beginning at 10 mg for 4 weeks, followed by 20 mg for 4 weeks, and then 30 mg for 4 weeks.
  Arms: Artesunate
Other: Placebo capsules — Placebo capsules
  Arms: Artesunate

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic progressive fibrotic lung disease resulting in increasing shortness of breath, cough, and low oxygen levels as a result of lung tissue scarring . This will be a single-center randomized, double-blinded, placebo-controlled study of 20 weeks including up to 4 weeks for screening, followed by 12 weeks of oral artesunate treatment across 3 dose levels (dose escalation every 4 weeks), and 4 weeks of a washout (follow-up) period in participants with Idiopathic Pulmonary Fibrosis (IPF). The primary objective of the study is to evaluate the safety and tolerability of artesunate at 3 dose levels, and to select the dose(s) to carry forward into additional clinical testing. The secondary objective includes exploring the blood biomarkers present in participants with IPF at baseline and to investigate how those biomarkers change following artesunate treatment. The exploratory objectives include assessing the changes in the K-BILD and Leicester cough questionnaire scores and change in pulmonary function after artesunate administration.

ELIGIBILITY:
Inclusion Criteria:

1. Participants, aged 40 years or older.
2. Diagnosis of IPF based upon ATS/ERS/JRS/ALAT 2018 guidelines (55).
3. FVC percent of predicted ≥ 40%; historical FVC for entry in the study is permitted if within 3 months of screening.
4. Diffusing capacity of lung for carbon monoxide (DLco) (hemoglobin-adjusted) ≥ 30%; historical DLco for entry in the study is permitted if within 3 months of screening.
5. Participants currently receiving treatment for IPF with nintedanib or pirfenidone are allowed, provided these drugs have been given at a stable dose for at least 6 weeks before the Screening visit (stable dose is defined as the highest dose tolerated by the participant during ≥ 6 weeks).
6. Female participants of childbearing potential (i.e., ovulating, premenopausal, and not surgically sterile) and all male participants with sexual partners of childbearing potential must use highly effective methods of birth control during their participation in the study and for 60 days after the last administration of study drug. Highly effective methods of birth control are defined as those with 99% or greater efficacy.
7. Participants must agree to abstain from egg or sperm donation through 60 days, after administration of the last dose of study drug.
8. Able to read and sign a written informed consent form (ICF).

Exclusion Criteria:

1. Receiving any nonapproved agent intended for treatment of fibrosis in IPF or Participation in other clinical trials.
2. Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, or sinusitis that can affect FVC measurement during screening.
3. Known acute IPF exacerbation or suspicion by the Investigator of such, within 3 months of screening.
4. The extent of emphysema is greater than the fibrotic changes on the most recent HRCT scan as determined by PI.
5. Any medical condition, not limited to cardiac, hepatic, renal disease or malignancy in recent months that will make the patients ineligible for the study, as deemed significant by PI.
6. Any of the following liver function test criteria above specified limits: total bilirubin >2× the upper limit of normal (ULN); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3× ULN; alkaline phosphatase > 2.5× ULN, pending PI's discretion.
7. Hemoglobin levels < 10.0 g/dL.
8. Pregnant or lactating females.
9. Likely to have lung transplantation during the study (being on transplantation list is acceptable).
10. Currently receiving and expected to remain on treatment during the study with: amodiaquine, and efavirenz, nevirapine and ritonavir.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience treatment-related adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mooney, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No